CLINICAL TRIAL: NCT07210450
Title: The Effect of Glutamine on Reducing Pulmonary Arterial Pressure in Non-transfusion-dependent Thalassemia Patients: a Single Blind Randomized Clinical Trial
Brief Title: Effect of L-Glutamine on Pulmonary Artery Pressure in Patients With Non-Transfusion-Dependent Thalassemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Rozita Gorzin, Pediatrician, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.MAZUMS.REC.1402.246
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Artery Pressure; Thalassemia; Non-transfusion Dependent Thalassemia
Keywords: L-glutamine; Non-transfusion Dependent Thalassemia; pulmonary artery pressure
MeSH Terms: conditions — Thalassemia | interventions — Glutamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Glutamine + Standard Care (Experimental): Participants in this arm will receive oral L-glutamine at a dose of 0.1 g/kg/day for 60 days, in addition to their routine standard care for non-transfusion-dependent thalassemia
  Interventions: Drug: L-glutamine
- Standard Care Alone (No Intervention): Standard care may include iron chelation therapy and/or hydroxyurea as prescribed by the treating physician.

INTERVENTIONS:
Drug: L-glutamine — Oral L-glutamine powder, administered at a dose of 0.1 g/kg/day for 60 days in adult patients with non-transfusion-dependent thalassemia (NTDT). The supplement is given in addition to each participant's standard care regimen (e.g., hydroxyurea or iron chelation therapy, as clinically indicated).
  Arms: L-Glutamine + Standard Care

SUMMARY:
The goal of this clinical trial is to learn whether L-glutamine can help lower pulmonary artery pressure in adults with non-transfusion-dependent thalassemia (NTDT).

The main questions it aims to answer are:

Does L-glutamine reduce pulmonary artery pressure after 60 days of treatment?

Is the effect of L-glutamine different from standard care alone?

Researchers will compare two groups:

Intervention group: Participants receive oral L-glutamine in addition to their standard treatment.

Control group: Participants continue with standard treatment only.

Participants will:

Take either L-glutamine (by mouth) or standard care for 60 days. Undergo echocardiography at the beginning and end of the study to measure pulmonary artery pressure.

Attend follow-up visits to monitor safety, adherence, and possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years), any sex.
* Diagnosis of non-transfusion-dependent β-thalassemia (NTDT).
* Pulmonary artery pressure (PAP) > 35 mmHg estimated by Doppler echocardiography at screening.
* Able and willing to provide written informed consent.
* On a stable standard-of-care regimen (e.g., chelation and/or hydroxyurea) per treating physician judgment.

Exclusion Criteria:

* Age <18 years.
* Refusal or inability to provide informed consent.
* Hepatic dysfunction: ALT >3× upper limit of normal.
* Renal dysfunction: serum creatinine >2× upper limit of normal.
* Known hypersensitivity to L-glutamine.
* Pregnancy or breastfeeding.
* Use of amino-acid/protein supplements within the past 3 months.
* History of other cardiac diseases associated with pulmonary hypertension (per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-09-27 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Artery Pressure (PAP) | Baseline to 60 days
  Pulmonary artery pressure (PAP) will be measured by Doppler echocardiography at baseline and at 60 days. The primary endpoint is the change in PAP (ΔPAP = Follow-up PAP - Baseline PAP) to assess whether L-glutamine reduces pulmonary artery pressure compared with standard care alone.

SECONDARY OUTCOMES:
Clinical Response Rate | 60 days
  Proportion of participants achieving either an absolute reduction in PAP ≥10 mmHg or a relative reduction ≥20% from baseline.
Safety and Tolerability of L-Glutamine | Baseline to 60 days
  Monitoring of adherence, adverse events, and treatment discontinuations related to L-glutamine supplementation.
Iron Load | Baseline to 60 days
  Association between change in pulmonary artery pressure (ΔPAP) and iron overload indices (Cardiac T2*, Liver T2*, and Liver Iron Concentration).

CONTACTS AND LOCATIONS:
Locations (1):
- Bu'Ali Sina Hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared because of the small sample size, the single-center design, and the need to protect patient privacy. Only aggregated results will be reported in publications or presentations.